CLINICAL TRIAL: NCT01365793
Title: Fluid Therapy and Cerebral Injury in Pediatric Diabetic Ketoacidosis
Brief Title: Randomized Control Trial of Fluid Therapy for Pediatric Diabetic Ketoacidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 230233; U01HD062417 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Cerebral Edema; Diabetic Ketoacidosis
Keywords: cerebral edema; diabetic ketoacidosis; pediatric diabetes; fluid therapy
MeSH Terms: conditions — Brain Edema; Diabetic Ketoacidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rapid rehydration using 0.45% saline replacement fluid (Experimental): This arm will involve more rapid intravenous fluid treatment which will include a second 10cc/Kg bolus of 0.9% saline and assume a 10% fluid deficit. 0.45% saline will be used as the replacement fluid for this arm.
  Interventions: Drug: 0.45% saline replacement fluid
- Rapid rehydration using 0.9% saline replacement fluid (Experimental): This arm will involve more rapid intravenous fluid treatment which will include a second 10cc/Kg bolus of 0.9% saline and assume a 10% fluid deficit. 0.9% saline will be used as the replacement fluid.
  Interventions: Drug: 0.9% saline replacement fluid
- Slower rehydration using 0.45% saline intravenous fluid (Experimental): This arm will involve slower rehydration (assumed 5% fluid deficit and no additional fluid bolus) with 0.45% saline used as the replacement fluid.
  Interventions: Drug: 0.45% saline intravenous fluid
- Slower rehydration using 0.9% saline intravenous fluid (Experimental): This arm will involve slower rehydration (assumed 5% fluid deficit and no additional fuid bolus) with 0.9% saline used as the replacement fluid.
  Interventions: Drug: 0.9% saline Intravenous fluid

INTERVENTIONS:
Drug: 0.45% saline replacement fluid — 10cc/Kg bolus of 0.9% saline followed by 0.45% saline used as the replacement fluid
  Arms: Rapid rehydration using 0.45% saline replacement fluid
Drug: 0.9% saline replacement fluid — 10cc/Kg bolus of 0.9% saline followed by 0.9% saline used as the replacement fluid.
  Arms: Rapid rehydration using 0.9% saline replacement fluid
Drug: 0.45% saline intravenous fluid — 0.45% saline fluid
  Arms: Slower rehydration using 0.45% saline intravenous fluid
Drug: 0.9% saline Intravenous fluid — 0.9% saline fluid
  Arms: Slower rehydration using 0.9% saline intravenous fluid

SUMMARY:
The investigators will conduct a randomized controlled trial comparing four different intravenous (IV) fluid treatment protocols for pediatric diabetic ketoacidosis (DKA). Two rates of rehydration will be compared; a more rapid rate and a slower rate. Within each of these two basic rehydration protocols, the investigators will vary the type of rehydration fluid used (0.9% saline or 0.45% saline). The investigators will compare the different treatments by conducting assessments of neurological injury, by measuring the frequency of significant cerebral edema, and by measuring long-term neurocognitive function.

These studies will allow us to determine whether variations in IV fluid treatment protocols affect acute neurological outcomes of DKA. Additionally, they will provide important data regarding the impact of DKA and DKA treatment on long-term neurocognitive function in children. In this way, the investigators hope to identify a more ideal fluid management strategy for children with DKA.

Previous studies have suggested that DKA may cause blood flow to the brain to be reduced and that brain injury might result from this reduction in blood flow and/or the effects of re-establishment of normal blood flow during DKA treatment with insulin and iv fluids. The investigators hypothesize that more rapidly re-establishing normal blood flow to the brain during DKA, by giving fluids more rapidly and using fluids with a higher sodium (salt) content, will help to minimize brain injury caused by DKA.

DETAILED DESCRIPTION:
These data will be compared to observational data from children with type 1 diabetes without DKA.

ELIGIBILITY:
Inclusion Criteria:

* must present or be transferred to a participating emergency department
* age less than 18 years
* diagnosis of DKA

  * serum glucose or fingerstick glucose concentration >300 mg/dL
  * venous pH < 7.25 OR serum bicarbonate concentration < 15 mmol/L.

Exclusion Criteria:

* patients with underlying neurological disorders or neurocognitive deficits which would affect either mental status testing during treatment or subsequent neurocognitive testing after recovery
* patients who present with concomitant alcohol or drug use, head trauma, meningitis or other conditions which might affect neurological function
* patients transferred to one of the participating emergency departments after initiation of DKA treatment other than one 10cc/kg intravenous bolus of 0.9% saline
* patients who are known to be pregnant at time of ED evaluation
* patients who have been enrolled in this study twice previously
* patients for whom the treating physician believed a specific fluid and electrolyte regimen was warranted
* patients for whom informed consent could not be obtained within 1 hour after completion of the initial fluid bolus, or within 2 hours from initiation of fluids, whichever is longer
* Patients who have been receiving IV fluids at a maintenance rate or greater (defined by the 4-2-1 rule) for more than two hours; OR
* Patients for whom it has been more than four hours since DKA therapy (IV fluids, IV bolus, or IV insulin) began; OR
* Patients who have been given hyperosmolar therapy (i.e. mannitol or 3% normal saline) prior to or since arriving at one of the participating PECARN emergency departments; OR
* Patients for whom the treating physician intends to immediately administer hyperosmolar therapy (i.e. mannitol or 3% normal saline); OR
* Patients whose baseline GCS is 11 or less.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1389 (Actual)
Dates: Start 2010-11; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Kuppermann, MD, MPH, Principal Investigator — University of California, Davis; Nicole S Glaser, MD, Principal Investigator — University of California, Davis
Locations (13):
- United States (13):
  - University of California, Davis, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University & St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hasbro Children's Hospital/Rhode Island Hospital, Providence, Rhode Island
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glaser NS, Ghetti S, Casper TC, Dean JM, Kuppermann N; Pediatric Emergency Care Applied Research Network (PECARN) DKA FLUID Study Group. Pediatric diabetic ketoacidosis, fluid therapy, and cerebral injury: the design of a factorial randomized controlled trial. Pediatr Diabetes. 2013 Sep;14(6):435-46. doi: 10.1111/pedi.12027. Epub 2013 Mar 13. PMID 23490311
- See also: Official website of the Pediatric Emergency Care Applied Research Network (PECARN), funded by HRSA/MCHB — http://www.pecarn.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapid Rehydration Using 0.45% Saline Replacement Fluid: This arm involved more rapid intravenous fluid treatment which included a second 10cc/Kg bolus of 0.9% saline and assumed a 10% fluid deficit. Intravenous fluids were infused to replace half of the estimated fluid deficit over 12 hours and the remaining half over the following 24 hours, in addition to maintenance fluids. 0.45% saline was used as the replacement fluid for this arm.
- Rapid Rehydration Using 0.9% Saline Replacement Fluid: This arm involved more rapid intravenous fluid treatment which included a second 10cc/Kg bolus of 0.9% saline and assumed a 10% fluid deficit. Intravenous fluids were infused to replace half of the estimated fluid deficit over 12 hours and the remaining half over the following 24 hours, in addition to maintenance fluids. 0.9% saline was used as the replacement fluid for this arm.
- Slower Rehydration Using 0.45% Saline Replacement Fluid: This arm involved slower rehydration (assumed 5% fluid deficit and no additional fluid bolus). Intravenous fluids were infused to replace the estimated deficit over 48 hours, in addition to maintenance fluids. 0.45% saline was used as the replacement fluid for this arm.
- Slower Rehydration Using 0.9% Saline Replacement Fluid: This arm involved slower rehydration (assumed 5% fluid deficit and no additional fluid bolus). Intravenous fluids were infused to replace the estimated deficit over 48 hours, in addition to maintenance fluids. 0.9% saline was used as the replacement fluid for this arm.
Period: Overall Study
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
Started | 344 | 351 | 345 | 349
Completed | 342 | 344 | 338 | 347
Not Completed | 2 | 7 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid | Total
Number analyzed (Participants) | 344 | 351 | 345 | 349 | 1389
Age, Customized [Count of Participants; unit: Participants]
  0 to less than 6 years old | 43 | 42 | 42 | 35 | 162
  6 to less than 18 years old | 301 | 309 | 303 | 314 | 1227
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 187 | 187 | 186 | 739
  Male | 165 | 164 | 158 | 163 | 650
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 235 | 232 | 247 | 243 | 957
  Race: Black or African American | 73 | 82 | 68 | 63 | 286
  Race: Other | 19 | 14 | 16 | 23 | 72
  Race: Unknown | 17 | 23 | 14 | 20 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 48 | 62 | 49 | 69 | 228
  Ethnicity: Not Hispanic or Latino, Other, or Unknown | 296 | 289 | 296 | 280 | 1161

OUTCOME MEASURES:

1. Primary Outcome: the Number of Participants With Glasgow Coma Score (GCS) < 14 Within the First 24 Hours of Treatment for Diabetic Ketoacidosis (DKA)
Description: The primary outcome is the binary indicator that a patient's GCS score drops below 14 (i.e. abnormal score) within the first 24 hours of treatment of DKA. There will be two treatment factors: sodium concentration of re-hydration fluids and rate of rehydration. These effects will be tested separately, using the Mantel-Haenszel chi-square test, stratified by hospital, and by the other main factor.
Time Frame: 24 hours
Population: Patients with a GCS of 14 or 15 at randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
Number analyzed (Participants) | 337 | 345 | 338 | 341
Participants | 10 | 11 | 11 | 16
Statistical Analysis 1: Comparison: Rapid Rehydration Using 0.45% Saline Replacement Fluid vs Rapid Rehydration Using 0.9% Saline Replacement Fluid vs Slower Rehydration Using 0.45% Saline Replacement Fluid vs Slower Rehydration Using 0.9% Saline Replacement Fluid; The study uses a factorial experimental design, and tests two null hypotheses. The first of these hypotheses - the frequency of GCS score declines to <14 is equal between the Rapid Rehydration and Slower Rehydration groups - is reported here. The analysis of the second hypothesis is reported below; Test type: Superiority — Each statistical test uses stratification to adjust for enrolling hospital, and the arm not being tested (e.g., the test for rapid vs slower rehydration is stratified by 0.45% and 0.9% Saline, and vice versa); p = 0.34, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance for each of the 2 p-values is 0.025, for an overall significance of 0.50
Statistical Analysis 2: Comparison: Rapid Rehydration Using 0.45% Saline Replacement Fluid vs Rapid Rehydration Using 0.9% Saline Replacement Fluid vs Slower Rehydration Using 0.45% Saline Replacement Fluid vs Slower Rehydration Using 0.9% Saline Replacement Fluid; The study uses a factorial experimental design, and tests the two null hypotheses. The second of these hypotheses - the frequency of GCS score declines to <14 is equal between the 0.45% Saline group and the 0.90% Saline group - is reported here. The analysis of the first hypothesis is reported above; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.43, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Frequency of Clinically Apparent Brain Injury
Description: Deterioration in neurological status requiring interventions such as hyperosmolar therapy or endotracheal intubation, or resulting in death. This outcome was determined by an adjudication committee.
Time Frame: 24 hours
Population: All randomized patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
Number analyzed (Participants) | 344 | 351 | 345 | 349
Participants | 2 | 2 | 5 | 3

3. Secondary Outcome: Hourly Improvement in Forward and Backward Digit Span Scores During DKA Treatment (Mean Difference Per Hour)
Description: The Digit Span subtest is adapted from the Wechsler Intelligence Scale for Children, 4th version (WISC-IV) and it assesses working memory. It consists of a Digit Span Forward task in which individuals are asked to repeat numbers in the same sequence as they were presented verbally and a Digit Span Backward task in which participants repeat the numbers in the reversed order to which they were heard. Each task yields a score ranging from 0 to 16. Higher scores represent better outcomes for this test. The trajectory of digit span scores during the course of the hospitalization was used to assess improvements in mental status and whether these varied systematically as a function of treatment protocol. Digit span measurements were collected every four hours during waking hours (7AM to 10PM). The measure analyzed is the average linear change in scores between enrollment and either 24-hours or DKA resolution, whichever occurred first.
Time Frame: 24 hours
Population: All randomized patients with digit span measured during DKA
Measure: Mean (Standard Error); unit: Digit Span Change per Hour
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
Number analyzed (Participants) | 344 | 351 | 345 | 349
Digit Span Change per Hour
  Digit span recall test Forward slope | 0.065 (0.010) | 0.058 (0.010) | 0.046 (0.010) | 0.039 (0.010)
  Digit span recall test Backward slope | 0.052 (0.009) | 0.053 (0.009) | 0.042 (0.009) | 0.043 (0.009)

4. Secondary Outcome: Mean Scores on Tests of Memory Capacity 3 Months After Recovery From DKA.
Description: Contextual memory was assessed via color and spatial-position tasks. Color-Task: black-ink items on a white square background were shown on a computer screen with a colored border. Subjects were asked to remember the item and the item's border color. Items were shown for 1 second, followed by a 1-second interval in which a fixation point was shown. Then, subjects were given a self-paced recognition test including studied drawings and new drawings shown in random order with no color border. Subjects determined if they had seen the drawing before. For recognized drawings, subjects reported the previously shown border color. Spatial-Position task: identical to the color task except that the items instead varied in their spatial position on the computer screen. The item-context association rate is the rate of correct item-color and item-spatial position recalled over the total of previously viewed items correctly recognized. Score range: 0-1 with higher scores indicating a better outcome.
Time Frame: 3 months
Population: All randomized subjects aged 6 years old and older with 3-month follow-up and successful completion of memory score tests, and d-prime (a measure of chance agreement) >0.50
Measure: Mean (Standard Deviation); unit: Item-context association rate
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
Number analyzed (Participants) | 175 | 184 | 178 | 176
Item-context association rate | 0.60 (0.14) | 0.60 (0.14) | 0.61 (0.14) | 0.60 (0.14)

5. Secondary Outcome: Intelligence Quotient (IQ) Testing
Description: IQ was assessed with the WASI (6-18 year olds) or WPPSI-III (3-5 year olds) at the 3 month follow-up visit. The Wechsler Abbreviated Scale of Intelligence (WASI) is a measure of IQ designed for individuals aged 6 to 89. The WASI includes four subtests; the Block Design and Matrix Reasoning tests measure Performance IQ, and the Vocabulary and Similarities tests measure Verbal IQ. Full scale IQ was computed from these scores and used for analyses. Scores typically vary from 75 to 135 with higher scores representing a better outcome.
Time Frame: 3 months
Population: All randomized subjects aged 3 years and older with 3-month follow-up and successful completion of IQ testing.
Measure: Mean (Standard Deviation); unit: IQ points
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
Number analyzed (Participants) | 187 | 201 | 191 | 189
IQ points | 102 (12) | 102 (13) | 102 (13) | 103 (13)

ADVERSE EVENTS:
Arm/Group | Rapid Rehydration Using 0.45% Saline Replacement Fluid | Rapid Rehydration Using 0.9% Saline Replacement Fluid | Slower Rehydration Using 0.45% Saline Replacement Fluid | Slower Rehydration Using 0.9% Saline Replacement Fluid
All-Cause Mortality (participants affected / at risk) | 1/342 | 0/344 | 0/338 | 0/347
Serious Adverse Events (participants affected / at risk) | 5/342 | 4/344 | 11/338 | 10/347
Other Adverse Events (participants affected / at risk) | 112/342 | 124/344 | 117/338 | 129/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Rehydration Using 0.45% Saline Replacement Fluid (N=342) | Rapid Rehydration Using 0.9% Saline Replacement Fluid (N=344) | Slower Rehydration Using 0.45% Saline Replacement Fluid (N=338) | Slower Rehydration Using 0.9% Saline Replacement Fluid (N=347)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2) | 2 (2) | 8 (8) | 7 (7)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Rehydration Using 0.45% Saline Replacement Fluid (N=342) | Rapid Rehydration Using 0.9% Saline Replacement Fluid (N=344) | Slower Rehydration Using 0.45% Saline Replacement Fluid (N=338) | Slower Rehydration Using 0.9% Saline Replacement Fluid (N=347)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nodal Rythm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 11 (11) | 7 (7) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2) | 5 (5)
Oesophageal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (4)
Catheter site inflammation (General disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Catheter site pain (General disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crying (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Infusion site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 8 (8) | 11 (11) | 8 (8) | 10 (10)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Candiduria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Otitits media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vuvlovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood chloride increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine phosphokinase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 4 (4)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood immunoglobulin A increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood ketone body increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood osmolarity decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood potassium decreased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coma scale abnormal (Investigations) | 0 (0) | 4 (4) | 1 (2) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave peaked (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary casts (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 3 (3) | 16 (16) | 4 (4) | 20 (20)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 4 (4) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 10 (10) | 9 (10) | 12 (13) | 15 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9) | 15 (15) | 8 (8) | 15 (16)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 5 (5) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 2 (2) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 29 (29) | 16 (16) | 23 (23) | 28 (31)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (5) | 5 (5) | 4 (4) | 6 (6)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (11) | 10 (10) | 9 (9)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Fluid infusion rates for this study represent the upper and lower ends of DKA protocols in use. Rates above or below this range were not evaluated. There were fewer patients with GCS decline to <14 than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No